CLINICAL TRIAL: NCT00133679
Title: Chronic Sildenafil for Severe Diaphragmatic Hernia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in clinical practice allowing chronic therapy at 6 weeks of age, incompatible with possibility of placebo beyond 6 weeks of age on study protocol
Sponsor: University of California, San Francisco (Other)
Collaborators: Children's Hospital Los Angeles (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23HL079922-01 (NIH)
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Hernia, Diaphragmatic; Hypertension, Pulmonary; Hypoplasia, Pulmonary
Keywords: Chronic lung disease; Nitric oxide; cyclic guanosine monophosphate; phosphodiesterase inhibitor
MeSH Terms: conditions — Hernia, Diaphragmatic; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sildenafil x 45 days
  Interventions: Drug: sildenafil
- 2 (Placebo Comparator): Placebo x 45 d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sildenafil — Sildenafil 0.5 mg/kg every 6 hours orally x 45 d
  Other Names: Viagra, Revatio
  Arms: 1
Drug: Placebo — Placebo suspension (equal volume to experimental drug) x 45 days
  Arms: 2

SUMMARY:
The purpose of this study is to test if sildenafil is effective in the treatment of infants with severe congenital diaphragmatic hernia (determined by the presence of prolonged pulmonary hypertension or prolonged oxygen supplementation on mechanical ventilation), as measured by the estimated pulmonary artery systolic pressure following treatment.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) is a condition characterized by pulmonary parenchymal and vascular hypoplasia. Severe CDH carries a high rate of mortality, and significant morbidity among survivors. This proposal is a randomized, blinded, placebo-controlled study designed to evaluate the efficacy and potential mechanisms of activity of sildenafil, a phosphodiesterase-5 inhibitor, for treatment of severe CDH. Infants who meet criteria at ≥10d of age predicting a poor outcome [death or chronic lung disease (CLD) severe enough to require hospital discharge on supplemental oxygen (O2)] will be eligible for the study. Infants whose parents consent for the study will undergo an initial echocardiogram to assess the degree of pulmonary hypertension. They will then begin either sildenafil or placebo therapy for a 45d course. A final echocardiogram will be performed after the experimental drug course is completed. The pulmonary arterial systolic pressure estimate during hyperoxic conditions will be compared between the sildenafil and placebo groups. Infants from either group who have severely elevated pulmonary arterial pressure (despite supplemental O2) will be considered for open-label sildenafil, which will continue after hospital discharge, depending on the results of a cardiac catheterization performed for clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Congenital diaphragmatic hernia
* 10-42 days (d) of age
* Significant illness severity as demonstrated by:
* Receiving assisted ventilation and

  * FiO2 >= 0.40 at 10-14d of age, or
  * FiO2 >= 0.40 for >=48hours at 15-27d of age, or
  * FiO2 >= 0.35 at 28-42d of age
* Or, need for extracorporeal support at >=10d of age
* Or, estimated pulmonary arterial or right ventricular systolic pressure of >= 2/3 systemic pressure at 14-42d of age

Exclusion Criteria:

* Structural congenital heart disease (other than patent ductus arteriosus or patent foramen ovale/atrial septal defect [ASD] or non-hemodynamically significant ventricular septal defect [VSD])
* Sildenafil contraindicated (until condition resolves):

  * Unable to absorb oral medication, or
  * Unstable systemic blood pressure, or
  * Receiving a drug that may interfere with sildenafil metabolism, or
  * Renal insufficiency
  * Hepatic insufficiency Previous use of sildenafil

Ages: 10 Days to 42 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2006-02; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta L Keller, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco Children's Hospital, San Francisco, California
  - Children's Memorial Hospital, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Groups:
- Sildenafil: Sildenafil x 45 days
  sildenafil: Sildenafil 0.5 mg/kg every 6 hours orally x 45 d
- Placebo: Placebo x 45 d
  Placebo: Placebo suspension (equal volume to experimental drug) x 45 days
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Estimated Systolic Pulmonary Arterial Pressure at Final Echocardiogram
Time Frame: 7 weeks
Population: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Systemic Levels of Vasoactive Substances at the Time of Final Echocardiogram
Time Frame: 7 weeks
Population: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Adverse Effects of Sildenafil Therapy
Time Frame: 2 years
Population: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Somatic Growth at 1 and 2 Years of Age
Time Frame: 2 years
Population: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Neurodevelopmental Outcome at 1 and 2 Years of Age
Time Frame: 2 years
Population: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Respiratory Status at 1 and 2 Years of Age
Time Frame: 2 years
Population: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Description: Study was terminated. All efforts to locate the data have been exhausted and data has been lost and/or destroyed.
Arm/Group | Sildenafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes